CLINICAL TRIAL: NCT05417282
Title: Safety and Tolerability of MW151 Administered With Whole-brain Radiotherapy in Patients With Intracranial Metastases
Brief Title: MW151 and Whole-brain Radiotherapy in Patients With Intracranial Metastases
Acronym: MW151-102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoChem Therapeutics, LLC (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Northwestern Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MW151-102; R44CA236382 (NIH)
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Cognitive Dysfunction, Cognitive Disorder
Keywords: MW151, MW01-2-151SRM, whole brain radiation therapy
MeSH Terms: conditions — Cognitive Dysfunction | interventions — 2-(4-(4-methyl-6-phenylpyridazin-3-yl)piperazin-1-yl)pyrimidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Safety and tolerability evaluation (Experimental): Part A: Open Label sentinel cohort 10 subjects will receive MW151 in an open label safety evaluation.
  Part B: Open Label 30 subjects will receive MW151.
  Interventions: Drug: MW151

INTERVENTIONS:
Drug: MW151 — Females: 20 mg MW151 daily (10 mg capsule BID), for 28 days; Males: 10 mg MW151 daily (10 mg capsule QD), for 28 days.
  Other Names: MW01-2-151SRM

SUMMARY:
HYPOTHESIS: MW151 intervention during whole-brain radiotherapy for intracranial metastases is safe and will mitigate neurocognitive decline.

RATIONALE: There is non-clinical evidence that MW151 reduces brain inflammation and improves neurocognitive outcomes in animal models of radiation therapy induced cognitive dysfunction, and in animal models of other CNS disorders.

PURPOSE: This feasibility trial will study whether MW151 mitigates neurocognitive decline following whole-brain radiotherapy in adult patients with intracranial metastases from solid tumors.

DETAILED DESCRIPTION:
In Part A, 10 subjects will receive MW151 in an open label evaluation. At least 5 of these subjects will be male. For each subject, safety and tolerability data for the first 24 hours will be reviewed prior to the continuation of dosing. Subjects will also be evaluated for safety during week 1, during week 2, and at week 4. Once the data from Part A have been reviewed by the Safety Monitoring Committee (SMC) for males and females, an additional 30 subjects will be recruited to Part B. These subjects will also receive open label MW-151.

In both parts A and B subjects will take study drug (males), or the first daily dose of study drug (females) before WBRT which will be administered once a day (3Gy), five days a week (Monday to Friday) for two weeks, for total of ten treatments and 30 Gy.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in the study only if all of the following criteria are met:

1. All patients must be willing to and have the capacity to give written informed consent and have signed and dated the informed consent form (ICF) in accordance with ICH and GCP guidelines, as an assurance that all participants understand the risks and benefits of the study
2. All patients must be able to speak and understand English proficiently
3. Histologically or cytologically confirmed diagnosis of a solid tumor malignancy within the past 5 years

   a. If the original histologic proof of malignancy is > 5 years, then pathological (i.e., more recent) confirmation is required (e.g., from a systemic metastasis or brain metastasis)
4. Intracranial metastases (either parenchymal brain metastases orleptomeningeal disease (LMD, also known as neoplastic meningitis, leptomeningeal carcinomatosis, or carcinomatous meningitis)) must be visible on contrast-enhanced MRI

Exclusion Criteria:

A subject will not be eligible for inclusion in the study if any of the following criteria are met:

1. Subject is lactating or is pregnant
2. Severe, active co-morbidity, defined as follows:

   1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
   2. Transmural myocardial infarction within the last 6 months
   3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
3. Intractable seizures while on adequate anticonvulsant therapy (i.e., more than one seizure per month for the past 2 months)
4. Clinically significant abnormalities in screening laboratory tests that would affect patient safety as determined by the principal investigator
5. History of psychiatric disorder requiring ongoing medical management
6. History of substance abuse including alcohol within past 5 years Appropriately prescribed medication for the treatment of pain or other symptoms related to the underlying malignancy is acceptable
7. Chronic kidney disease defined as the presence of significant proteinuria on urinalysis and/or eGFR of <60mL/min, as calculated by the clinical site laboratory
8. Inability to follow the instructions or an unwillingness to cooperate with study procedures
9. Known allergy to any component of MW151 as described in investigator's brochure
10. Received treatment with and/or planned treatment with systemic chemotherapy within 3 days prior, during, or for at least 3 days after completion of whole-brain radiotherapy. Concurrent immunotherapy is permitted
11. Prior whole-brain radiotherapy
12. Use of chronic short-acting benzodiazepine
13. Use of chronic NSAID or steroid therapies for chronic inflammatory diseases within 3 days prior to dosing and during the course of the study drug dosing. Use of aspirin for cardiac prophylaxis is acceptable. Use of any other NSAID's or steroids should be reviewed by sponsor, approved and approval documented.
14. Any reason or opinion of the investigator that would prevent the subject from participation in the study
15. Currently receiving treatment with and/or planned treatment with Memantine HCl or combination drugs containing Memantine HCl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28 days
  To assess the safety and tolerability of oral administration of MW151 in adult patients with brain metastases.

SECONDARY OUTCOMES:
Reduction in cognitive deterioration | 6 months
  To determine if the addition of MW151 to WBRT standard of care treatment will show a trend towards reduction in cognitive deterioration in patients with brain metastases from solid tumors, as measured by standardized NCF tests.
Anti-inflammatory effects | 6 months
  To determine if the addition of MW151 to WBRT will have an impact on plasma levels of proinflammatory cytokines (PIC).
Progression-free survival and overall survival | 6 months
  To evaluate intracranial progression-free survival and overall survival following the addition of MW151 to WBRT standard of care treatment for patients with brain metastases.
Exploratory objective: brain age analysis in patiens undergoing whole-brain radiotherapy plus MW151 | 6 months
  To correlate the difference between brain age over time with neurocognitive function following whole-brain radiotherapy plus MW151 using SBDL (Surface-Based Deep Learning) brain age prediction.

CONTACTS AND LOCATIONS:
Overall Officials: Vinai Gondi, MD, Principal Investigator — Northwestern Medicine
Locations (1):
- Northwestern Memorial HealthCare, Central DuPage Hospital, Warrenville Cancer Center, Winfield, Illinois, United States

IPD SHARING:
Plan to Share IPD: No